CLINICAL TRIAL: NCT06227715
Title: Non-Carious Cervical Lesions Restorations Using Different Modes of Universal Adhesive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Hatice Tepe, Lecturer, Eskisehir Osmangazi University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 80558721/G-109
Record Dates: First submitted 2023-12-21; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Tooth Wear
Keywords: nccl; universal bond; acid etching; selective etching
MeSH Terms: conditions — Tooth Wear

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- selective etch (Other): In SLE mode, only enamel margin was etched for 15 seconds, washed for 15 seconds and dried, and the adhesive was applied to the dentin and enamel by rubbing for 20 seconds.
  Interventions: Other: universal adhesive
- Total etch (Other): Each mode of the universal adhesive used in the mouth of each of the patients evaluated was applied to at least two teeth. In accordance with the recommendations of the manufacturer; in TE mode, enamel and dentin were etched with 37% orthophosphoric acid for 15 seconds, washed for 15 seconds, and after air-drying, the adhesive was applied to enamel and dentin by rubbing for 20 seconds.
  Interventions: Other: universal adhesive
- self etch (Other): In SE mode, the adhesive was applied to the dentin and enamel by rubbing for 20 seconds.
  Interventions: Other: universal adhesive

INTERVENTIONS:
Other: universal adhesive

SUMMARY:
Objectives: To evaluate the 36-month clinical performance of Single Bond Universal Adhesive (SBU; 3M ESPE, Germany) in non-carious cervical lesions (NCCLs) using different modes adhesion approaches according to the FDI criteria.

Material and methods: SBU Adhesive was applied in 252 NCCLs of 25 patients using different modes adhesion approaches: Self-etch (SE), selective-enamel-etching (SLE), total-etch (TE). All lesions were restored with nanohybrid resin composite. Restorations were evaluated at baseline, 6th, 12th, 18th, and 36th month using the FDI criteria. IBM SPSS Statistics for Windows, Version 24.0. program was used in the analysis. Differences between SE, SLE and TE groups were tested using Kruskal Wallis test. A value of p<0.05 was accepted as a criterion for statistical significance.

DETAILED DESCRIPTION:
Study Design Non-Interventional Clinical Research Ethics Committee (80558721/G-109) approved the study. All participants were informed of the study and consent forms were obtained. The experimental design adhered to the Consolidated Standards of Reporting Trials (CONSORT) statements. For this retrospective study, between May 2015 and July 2015, 102 patients who were diagnosed with non-carious cervical lesion and had their restoration completed in Faculty of Dentistry by single operative dentist. 25 volunteers (10-females, 15-males) with the ages ranging from 35 to 72, 252 restorations were selected for this study according to predetermined criteria (table 1).

Sample Size Calculation G* Power statistical software was used to calculate the sample size. For an effect size (Cohen 'D Effect Size) difference of 0.30 between the groups with 99% power, DF=2 and an alpha error of 5%, at least 238 restorations were needed.

Patient Selection Adults who achieved the inclusion/exclusion criteria and required restoration of at least one notch shaped NCCL were included in the study. Inclusion criteria were the presence of at least 20 teeth and 6 NCCL, the absence of common caries, and the use of universal adhesive and nanohybrid resin composite. Candidates with poor oral hygiene, acute or chronic periodontal disease, xerostomia, and malocclusion were excluded.

The patient forms, in which the identity information of the patients participating in the study and the size of the lesion in the restored teeth, the type and mode of adhesive used in the restoration, and the restorative material were recorded, were reviewed and the necessary tooth groupings were made following the recorded data.

Application Procedure of Restorations The NCCL dimensions in millimeters (height and width) were determined with a digital caliper. Prior to the restoration procedures, a pumice stone and water were used for prophylactic purposes, then the dentin was abraded and beveled to the enamel surface (1-2 mm). Before the restoration of the lesions, isolation was achieved with the use of retraction cord (Ultrapak, Ultradent Products, USA) and cotton rolls. Three different application modes of the universal dentin bonding (Single Bond Universal, 3M ESPE, Germany) adhesive were applied in the restoration of the teeth (table 2). These are TE, in which both dentin and enamel are etched, SLE, in which only enamel is etched, and SE, in which only the adhesive is applied. Each mode of the universal adhesive used in the mouth of each of the patients evaluated was applied to at least two teeth. In accordance with the recommendations of the manufacturer; in TE mode, enamel and dentin were etched with 37% orthophosphoric acid for 15 seconds, washed for 15 seconds, and after air-drying, the adhesive was applied to enamel and dentin by rubbing for 20 seconds. In SLE mode, only enamel margin was etched for 15 seconds, washed for 15 seconds and dried, and the adhesive was applied to the dentin and enamel by rubbing for 20 seconds. In SE mode, the adhesive was applied to the dentin and enamel by rubbing for 20 seconds. After the adhesive was applied in all modes, it was dried for 5 seconds gently and polymerized 10 seconds using a curing light (SmartLite Focus, Dentsply Sirona, USA). Afterwards, all of them were restored with the same nanohybrid resin composite (Filtek Z550, 3M ESPE, USA) in accordance with the layering technique. Restorations were completed by polishing under water cooling with fine diamond burs (GZ Instrumente, Austria) and polishing discs (Soflex Finishing and Polishing Disc, 3M ESPE, USA).

Assessment of Restorations At the 1st, 6th, 12th, 18th, and 36th month, the restorations were evaluated based on the FDI criteria and the results were recorded on the clinical research follow-up form. Two calibrated experienced dentists evaluated the restorations without knowing which adhesive technique was used on which patient, except for the treating dentist, using a mirror and sond under reflector light.

Restorations were evaluated marginal staining, fracture of material and retention, marginal adaptation, post-operative sensitivity and vitality, recurrence of caries, erosion and abfraction, tooth integrity according to the FDI criteria. According to the FDI criteria, these variables were ranked as follows: clinically very good (1), clinically good (2), clinically satisfactory (3), clinically unsatisfactory (4), and clinically poor (5). In accordance with these criteria, values of 1,2 and 3 are clinically acceptable, while 4 and 5 are considered clinically not acceptable.16 The difference between the adhesive modes and the time-dependent variation within each mode were evaluated. Among the evaluated restorations, those with retention loss were evaluated only according to the retention loss criteria and scored with 5 and were not evaluated in terms of other criteria. Restorations that were unsuccessful due to either loss of retention or irreparable secondary caries were replaced with new composite resin restorations. These new restorations were then excluded from the study for further evaluation.

Statistical Analysis Descriptive statistics were used to present the frequency distributions. Shapiro Wilk's test was performed to evaluate the normality of data distribution and it was seen that data were not normally distributed. Differences between SE, SLE and TE groups were tested using Kruskal Wallis test. The was used to compare the groups at baseline, 6, 12, 18 and 36 months. To compare the data in marginal staining, fracture of material and retention, marginal adaptation, post-operative sensitivity and vitality, recurrence of caries, erosion and abfraction, tooth integrity within each group by time, further analyses were carried out using the K Releated Samples and Wilcoxon tests. IBM SPSS Statistics for Windows, Version 24.0. (Armonk, NY: IBM Corp., USA) program was used in the analysis. A value of p<0.05 was accepted as a criterion for statistical significance.

ELIGIBILITY:
Inclusion Criteria

* At least 20 teeth and 6 NCCL
* The absence of common caries
* The use of universal adhesive and nanohybrid resin composite

Exclusion Criteria

* Candidates with poor oral hygiene
* Acute or chronic periodontal disease
* Xerostomia,
* Malocclusion were excluded.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-04-28 (Actual); Primary Completion 2018-10-28 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Non-Carious Cervical Lesions Restorations Using Different Modes of Universal Adhesive | 6, 12, 18, 36, 60 month
  Restorations were evaluated marginal staining, fracture of material and retention, marginal adaptation, post-operative sensitivity and vitality, recurrence of caries, erosion and abfraction, tooth integrity according to the FDI criteria.
  Clinically excellent/very good (1) Clinically good (after polishing very good) (2) Clinically sufficient/satisfactory (minor shortcomings, no unacceptable effects but not adjustable w/o damage to the tooth) (3) Clinically unsatis- factory (but reparable) (4) Clinically poor (replacement necessary) (5)

REFERENCES:
- [Derived] Tepe H, Celiksoz O, Yaman BC. Clinical evaluation of single bond universal adhesive in non-carious cervical lesions: a 36-month retrospective study. Clin Oral Investig. 2024 Dec 28;29(1):33. doi: 10.1007/s00784-024-06126-y. PMID 39731636
- See also: FDI Criteria for dental restorations — https://link.springer.com/article/10.1007/s00784-010-0432-8